CLINICAL TRIAL: NCT00054418
Title: A Phase III Randomized, Placebo-Controlled, Double-Blind Trial Of Risedronate (Actonel) For Prevention Of Bone Loss In Premenopausal Women Undergoing Chemotherapy For Primary Breast Carcinoma
Brief Title: Risedronate in Preventing Bone Loss in Premenopausal Women Receiving Chemotherapy for Primary Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N02C1; NCI-2012-02515 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000270449 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: osteoporosis; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Calcium Carbonate; Vitamin D; Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- calcium carbonate, vitamin D and risedronate (Experimental): Patients receive calcium carbonate 600 mg daily, vitamin D 400 U daily and risedronate 35 mg weekly.
  Interventions: Dietary Supplement: calcium carbonate; Dietary Supplement: vitamin D; Drug: risedronate sodium
- calcium carbonate, vitamin D and placebo (Placebo Comparator): Patients receive calcium carbonate 600 mg daily, vitamin D 400 U daily and placebo weekly.
  Interventions: Dietary Supplement: calcium carbonate; Dietary Supplement: vitamin D; Other: placebo

INTERVENTIONS:
Dietary Supplement: calcium carbonate — calcium 600 mg daily administered orally for one year
Dietary Supplement: vitamin D — vitamin D 400 U daily administered orally for one year
Drug: risedronate sodium — risedronate 35 mg weekly administered orally
  Arms: calcium carbonate, vitamin D and risedronate
Other: placebo — placebo tablet weekly administered orally for one year
  Arms: calcium carbonate, vitamin D and placebo

SUMMARY:
RATIONALE: Preventing bone loss in patients who are receiving chemotherapy for breast cancer may decrease the risk of fractures and may help patients live more comfortably. It is not yet known whether calcium is more effective with or without risedronate in preventing bone loss.

PURPOSE: This randomized phase III trial is studying two forms of calcium with or without risedronate to compare how well they work in preventing bone loss in premenopausal women who are receiving chemotherapy for primary stage I, stage II, stage IIIA, or stage IIIB breast cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a randomized, placebo-controlled, double-blind study. Patients are stratified according to planned tamoxifen therapy (yes vs no vs undecided), planned taxane therapy (yes vs no vs undecided), time from last menses (1-3 months vs longer than 3 months to 6 months), and age (under 40 vs 40 to 49 vs 50 and over). Patients are randomized to 1 of 2 treatment arms. In both arms, treatment begins during the first month of chemotherapy and continues for 1 year in the absence of unacceptable toxicity. For more information regarding the treatment arms, please see the "Arms" section below. Questionnaires about cessation of menses, ovarian failure, and menopausal symptoms are completed at baseline, monthly during chemotherapy, at 6 months, and then at 1 and 2 years.

Patients are followed for 1 year. A summary of study goals is listed below.

Goals:

1. To evaluate the effectiveness of risedronate at a weekly oral dose of 35 mg versus placebo in the prevention of bone loss in premenopausal women undergoing adjuvant or neoadjuvant chemotherapy for primary breast cancer.
2. To evaluate the degree of bone loss over one year in premenopausal women undergoing adjuvant chemotherapy for primary breast cancer according to menopausal status at one year after therapy begins.
3. To evaluate the relationship of current climacteric symptoms, menstrual and reproductive history, and chemotherapy regimen with ovarian failure (permanent cessation of menses) in premenopausal women undergoing adjuvant or neoadjuvant chemotherapy for primary breast cancer.
4. To evaluate the relationship of baseline serum estradiol levels with ovarian failure in premenopausal women undergoing adjuvant or neoadjuvant chemotherapy for primary breast cancer.

ELIGIBILITY:
1. Required Characteristics

   1. Premenopausal women

      * ≤ 6 months since last menstrual period
      * no prior bilateral oophorectomy
      * not on estrogen replacement therapy
      * if TAH is performed, with at least one intact ovary, or if > 3 months since last menstrual period, then patients must have premenopausal estrogen levels ≤ 1 month of study entry
   2. Scheduled to undergo adjuvant or neoadjuvant chemotherapy for primary breast cancer (stages I-IIIB)
   3. ≥ 18 years of age
   4. ECOG performance status (PS) 0 or 1
2. Contraindications

   1. Hypercalcemia (calcium level > 1mg/dL above UNL ≤ 6 months
   2. Hypocalcemia (calcium level > 0.5 mg/dL below UNL ≤ 6 months
   3. Inability to stand or sit upright for at least 30 minutes
   4. Known swallowing disorder
   5. Bone mineral density T score of ≤ - 2.0 at the hip or lumbar spine

      * a patient with a T score of - 2.1 is ineligible
      * a patient with a T score of - 1.9 is eligible
   6. History of vertebral compression fracture

      * Exception: traumatic fracture of the coccyx would not exclude a patient from participation
   7. Corticosteroids at doses > 5 mg daily of prednison or equivalent for > 2 weeks in the past 6 months
   8. Previous treatment with bisphosphonates
   9. Diseases affecting bone metabolism (hyperthyroidism, hyperparathyroidism, and hypercortisolism)
   10. History of severe renal impairment or creatinine > 2.0 mg/dL
   11. Malabsorption syndrome
   12. Estrogen replacement therapy
   13. Oral contraceptive use
   14. Prior bilateral oophorectomy
   15. Pregnant women

       * Nursing women
       * Women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, injections, intrauterine device [IUD], surgical sterilization, abstinence, etc.)
       * This study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown
   16. Dental extraction, root canal, or implants ≤ 3 months prior to registration or planned during study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2003-03; Primary Completion 2007-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Average intra-patient change in lumbar spine (L2-L4, PA) bone mineral density (BMD) from baseline to one year after study entry | 1 year post study entry

SECONDARY OUTCOMES:
Average intra-patient change in femoral neck and total hip BMD from baseline to one year after study entry | 1 year post study entry
Incidence of osteopenia in the risedronate vs placebo groups at one year after study entry | 1 year post study entry
Incidence of osteoporosis in the risedronate vs placebo groups at one year after study entry | 1 year post study entry
Incidence of a 5% difference in intra-patient BMD scores at baseline | Baseline
Serum and urine N-telopeptide and serum alkaline phosphatase at baseline and 6 months | Up to 6 months
Frequency and severity of toxicity as measured by NCI CTC version 2.0 | Up to 1 year post study treatment
Menopausal symptoms as measured by the Greene Climacteric Scale (GCS) at baseline, monthly during chemotherapy, at 6 months, 1 year, and 2 years after study entry | Up to 2 years post study entry
Association of baseline serum estradiol levels with permanent cessation of menses | Baseline
Relationship between the subscales of the GCS (psychological, vasomotor, somatic and sexual) with type of chemotherapy, duration of chemotherapy, and menstrual cycle changes | Up to 2 years post study entry

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Hines, MD, Study Chair — Mayo Clinic
Locations (199):
- United States (198):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thorton, Colorado
  - Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, P. C., Ames, Iowa
  - Bettendorf, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Alegent Health Community Memorial Hospital, Missouri Valley, Iowa
  - Burgess Health Center, Onawa, Iowa
  - Ottumwa Regional Health Center Cancer Center, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates at June E. Nylen Cancer Center, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, P.A. - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, P.A. - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, P.A. - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, P.A. - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, P.A. - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, P.A. - Salina, Salina, Kansas
  - Cancer Center of Kansas, P.A. - Wellington, Wellington, Kansas
  - Associates in Womens Health, P.A. - North Review, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Winfield, Winfield, Kansas
  - Ochsner Clinic of Baton Rouge, Baton Rouge, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, P.C., Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Immanuel St. Joseph's Clinic, Mankato, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Hattiesburg Clinic, P.A., Hattiesburg, Mississippi
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine Associates of Bozeman, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - St. Elizabeth Regional Medical Center, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Toledo Surgical Specialists, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, P. C., Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Hines SL, Mincey BA, Sloan JA, Thomas SP, Chottiner E, Loprinzi CL, Carlson MD, Atherton PJ, Salim M, Perez EA. Phase III randomized, placebo-controlled, double-blind trial of risedronate for the prevention of bone loss in premenopausal women undergoing chemotherapy for primary breast cancer. J Clin Oncol. 2009 Mar 1;27(7):1047-53. doi: 10.1200/JCO.2008.19.1783. Epub 2008 Dec 15. PMID 19075260
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716